CLINICAL TRIAL: NCT00848679
Title: Investigating the Novel Observation of Right-left Difference in Uterine Artery Vascular Resistance in Pre-eclampsia: A Double-blinded, Randomized, Placebo-controlled Study to Assess the Dose-dependent Effect of Epidural Lidocaine on Right-left Uterine Artery Blood Flow Differences in Pre-eclampsia, With Healthy Term Pregnant and Non-pregnant Controls
Brief Title: Investigating the Novel Observation of Right-left Difference in Uterine Artery Vascular Resistance in Pre-eclampsia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACET3-ginosar-HMO-CTIL
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2009-02

CONDITIONS: Pre-eclampsia
Keywords: Pre-eclampsia; Pregnancy; Uteroplacental blood flow; Epidural; Anesthesia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epidural lidocaine (Active Comparator): 30 women to receive 5 x 5mL boluses of epidural lidocaine 2%. 10 pre-eclampsia, 10 term pregnancy, 10 non-pregnant.
  Interventions: Drug: Epidural lidocaine; Drug: Epidural lidocaine 2%
- Epidural saline (Placebo Comparator): 30 women to receive 5 x 5 mL boluses of epidural saline. 10 pre-eclamptics, 10 normal term pregnancy, 10 non-pregnant
  Interventions: Drug: Epidural lidocaine; Drug: Epidural lidocaine 2%

INTERVENTIONS:
Drug: Epidural lidocaine — Epidural 2% lidocaine, administered in 5mL incremental boluses. Looking at dose-response effect.
Drug: Epidural lidocaine 2% — 5 x 5ml boluses of either epidural lidocaine 2% or epidural saline

SUMMARY:
The investigators previously demonstrated that epidural ropivacaine reduces uterine artery vascular resistance in a dose dependent manner in pre-eclampsia. The investigators also noted a marked right-left difference in vascular resistance between paired uterine arteries, which was almost completely abolished following epidural ropivacaine. However, this novel observation was not a stated outcome variable before the study began. This study assesses right-left difference in vascular resistance between paired uterine arteries as a primary end-point, assesses the dose-response effect of epidural lidocaine and compares the effect observed in pre-eclampsia with that in two control populations (term normal pregnancy and non-pregnant controls).

ELIGIBILITY:
Inclusion Criteria:

* Pre-eclampsia patients and normal pregnancy controls scheduled to receive epidural catheterization for induction of labor or Cesarean delivery. Non-pregnant controls receiving epidural catheterization for elective surgery. Pre-eclampsia group:

  1. gestational age between 35 to 40 completed weeks
  2. uterine artery notching OR evidence of reduced uterine artery blood flow
  3. resting systolic pressure > 140mmHg or diastolic pressure > 90mmHg measured twice at least 6 hours apart
  4. proteinuria (at least 0•1 g/l in two random samples at least 6 hours apart or at least 0•3g in a 24 hour collection).
* Normal pregnancy control group:

  1. gestational age between 35 to 40 completed weeks
  2. absence of other inclusion factors for the pre-eclampsia group. Non-pregnant control group: Non-pregnant women of reproductive age.

Exclusion Criteria:

* Active labor, resting blood pressure ≥ 160/110 (recorded on at least two occasions 6 hours apart), coagulopathy or other contraindications for epidural catheterization, abnormal fetal heart tracing, known fetal anomaly, intrauterine infection, placental anomalies, twins, and refusal of consent.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2009-10 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Uterine artery pulsatility index (by Doppler ultrasound). Specifically the right-left uterine artery difference. | 15min after each dose - on a dose--response curve

SECONDARY OUTCOMES:
Uterine artery pulsatility index (worse vessel) | 15 min after dose

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Hebrew University Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Ginosar Y, Nadjari M, Hoffman A, Firman N, Davidson EM, Weiniger CF, Rosen L, Weissman C, Elchalal U; ACET study group. Antepartum continuous epidural ropivacaine therapy reduces uterine artery vascular resistance in pre-eclampsia: a randomized, dose-ranging, placebo-controlled study. Br J Anaesth. 2009 Mar;102(3):369-78. doi: 10.1093/bja/aen402. Epub 2009 Jan 27. PMID 19176534